CLINICAL TRIAL: NCT04849637
Title: Virgin Coconut Oil as Adjunctive Therapy for Hospitalized COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Philippines (Other)
Collaborators: Philippine Coconut Authority (Unknown); Philippine Council for Health Research & Development (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPMREB 2020-306-01
Record Dates: First submitted 2021-03-19; First posted 2021-04-19 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: virgin coconut oil; COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care plus adjunctive virgin coconut oil supplementation (Experimental): Standard of care plus virgin coconut oil
  Interventions: Drug: Virgin Coconut Oil
- COVID-19 Standard of care treatment (No Intervention): Standard of care

INTERVENTIONS:
Drug: Virgin Coconut Oil — Oral supplementation of virgin coconut oil to COVID-19 patients
  Other Names: VCO
  Arms: Standard of care plus adjunctive virgin coconut oil supplementation

SUMMARY:
This is a research that will investigate the safety and efficacy of virgin coconut oil (VCO) as an adjunctive therapy for Coronavirus Disease 2019 (COVID-19)

DETAILED DESCRIPTION:
This study will be a randomized controlled trial among hospitalized COVID-19 patients, aged 18 years old and above, admitted at the Philippine General hospital. Patients will be grouped into the following:

1. Group receiving standard of care
2. Group receiving standard of care plus virgin coconut oil (15ml, 3x/day for 2 weeks) as adjunctive therapy.

Patients will be observed as regards to primary outcomes such as recovery/resolution of symptoms and duration of hospital stay

ELIGIBILITY:
Inclusion Criteria:

* symptomatic and asymptomatic COVID-19 hospitalized patients
* has laboratory-confirmed illness during the time of recruitment
* able to take food and medicines enterally

Exclusion Criteria:

* uncontrolled or newly diagnosed diabetes mellitus
* with chronic heart disease
* having elevated lipid profile at baseline (admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-04-09 (Estimated); Study Completion 2022-04-09 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | Two weeks
  To determine if the VCO intervention can lessen the duration of stay in the hospital by at least 2 days
Time to recovery/resolution of symptoms | Two weeks
  Patient will be assessed based on the following secondary outcome: time interval before ventilation, ICU and negative results on PCR swab test

SECONDARY OUTCOMES:
Time to first receipt of ventilation and admission to intensive care unit | Two weeks
  monitor the duration by which symptoms progress to a point where patient may need intensive care unit admission and/or use of ventilation machine after onsent of VCO administration
IL-6 levels (pg/mL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
Ferritin levels (ng/mL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
CRP levels (mg/dL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
LDH levels (mg/dL0 | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
TNF-Alpha levels (pg/mL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
Interferon-gamma levels (pg/mL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
Monocyte chemoattractant protein levels (pg/mL) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
Immunoglobulin levels (mg/L) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database
CD4+ counts (cells/L) | Two weeks
  Peripheral blood (at most 5mL) will be collected from each patient at baseline, and every week thereafter until the end of study participation for secondary outcome emasurement (CD4+ cells). Blood extraction will coincide with blood collection for routine diagnostic workup of the patient. Laboratory results of other outcome parameters (ie IL6, CRP, ferritin, LDH) will be extracted from patient medical records (as aprt of routine work-up) or from patient database

OTHER OUTCOMES:
Negative test result for COVID by RT-PCR | Two weeks
  Negative test result for COVID by RT-PCR (within 3 days after the two week administration of VCO)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa M Alejandria, MD, Principal Investigator — UP Manila; Leslie Michelle M Dalmacio, PhD, Principal Investigator — UP Manila
Locations (1):
- Philippine General Hospital, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No